CLINICAL TRIAL: NCT00563043
Title: Pattern Scan Laser System vs Regular Photocoagulation System: Changes in Electroretinograms and Contrast Sensitivity Post Treatment.
Brief Title: Changes in Electroretinogram and Contrast Sensitivity After PASCAL Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Asociacion para evitar la ceguera en mexico, apec
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PASCAL002
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non Proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy
Keywords: Pattern Scan Laser.; Photocoagulation.; Diabetic retinopathy treatment.; Laser treatment.; Electroretinogram.; a wave.; b wave.; Implicit time.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PASCAL laser treatment — Patterns Scan Laser treatment in patients with PDR.

SUMMARY:
Laser photocoagulation has become the treatment of choice in PDR. Laser photocoagulation has become the treatment of choice in PDR. The aim is to destroy a substantial portion of the peripheral retina in order to reduce the angiogenic stimulus (decrease the difference between oxygen demand and the administration). Their effectiveness is determined by the extent of destruction of the retina (2.4).

DETAILED DESCRIPTION:
Introduction:

The concept of retinal photocoagulation was introduced by Meyer-Schwickerath for treatment of diabetic retinopathy in the 50s (1, 6). The first successfully used laser was the arc xenon laser (polychromatic, inefficient, and hard to handle). Then the ruby and argon laser appeared (with mayor improvements in design and management). The modern era of photocoagulation as we know it began in the late 70s.

With these available technologies, the focal photocoagulation, the panretinal photocoagulation and the grid photocoagulation were developed. Witch proved effective for the treatment of severe non-proliferative diabetic retinopathy, proliferative diabetic retinopathy in different multicenter studies (ETDRS, DRS) (1.6).

Patients usually receive from 1200 to 1500 laser shots in 2 to 4 sessions lasting from 10 to 20 minutes, during 2 to 4 weeks. The procedure can be time consuming, tedious and painful.

Until now little has changed in the overall design of lasers of 30 years ago. The differences are the introduction of fibre optics and air-based cooling systems. These innovations do not have any impact on the way in which the treatment or the success.

Early efforts to improve photocoagulation included complex recognition systems and eye tracking to try to manage a fully automated process. That required a preview image of the retina. Attempts were also made to determine the appropriate dose of energy for getting the job done. The complexity of these systems prevented their clinical use (1).

The PASCAL is a system of semiautomatic pattern laser, which allows much faster processing, accuracy and control of treatment by a doctor at all times. The difference with the regular laser systems is that PASCAL manages a dual frequency Nd: YAG that works at a wavelength of 532nm, which is capable of firing a single shot from up to 56 shots in pre patterns (1x1, 2 x2, 3x3, 4x4, 5x5). By using time exposures of between 10 and 20 ms, you can make multiple shots at the same time that a shot with conventional laser is done (100 ms). These short pulses allow energy laser focus better in the tissues, produces less pain, Reduce the heat delivered to the choroid, and less diffusion of heat with the subsequent less damage to surrounding tissues (1).

The first study was published in the Retina 2006, by Blumenkanz, Palanker, Marcelino, et al. In which describe their use in rabbit's retinas. In which compared the effect of a number of pulses of different durations and powers. They applied exposition of 10, 20, 50 and 100 ms. The study found that at lower exposure time is required energy of 2 to 3 times more to produce the same effect, but the pulse had less energy. As they increased the exposure time, les power was needed, but the pulsed had also more energy. As the energy increased the shots was less homogeneous, less localized and changes in the final size (110-170micm) (1).

ERG: It reflects the activity of the retina in "mass". In studies of the effect of photocoagulation on the activity of the retina, it have typically been used the amplitude of them a and b wave as criteria of tissue destruction. But there is no consistency among the various studies that have already reported variations of 10 to 95% in the amplitude (especially in wave b) due to the variability in the length of effective ablation of the retina. Others suggest that a wave to be smaller than the b, showing an injury in the primary layer of photoreceptors. Others say that the decline was equal in both waves. But something we all conclude is that the response in the ERG is reduced more than expected based in the coagulated area. But when it is higher, the fall in the ERG is more than what was expected (60% of destruction = 80% decrease of ERG). An average photocoagulation destroys about 40% of the retina approximately (5).

The destruction of the peripheral retina decreases the ERG response, besides laser affect regions of adjacent tissue, causing deterioration in the transmission of signals from the photoreceptors in the proximal retina. What explains the previous reports of large decrease in amplitude on the basis of the area coagulated (2). The laser energy is absorbed by the RPE cells, and the adjacent layer of photoreceptors. What also produces external injury to the retina so you can also observe an increase in the implicit time (3).

A few years ago changing arc xenon to argon marked a difference in the amount of burned retina and decrease in the implicit time and amplitudes of the waves (5).

Macular Edema: Is recognized as a potential adverse effect of panretinal photocoagulation. Witch may transitory or permanent decrease the visual acuity of the patient. Approximately 60% of photocoagulated patients show an increase in the foveal thickness. Despite the fact that it has been said that a change of the self-distribution of blood flow is responsible for this increase in the thickness, today it is believed that these changes are due to post-laser inflammation. Despite that it is performed outside of the vascular arches; it is generally formed by those within.

The inflammation factors, in addition to the direct effect that is exercised on intracellular unions have shown themselves capable of producing a change in the barrier mediated leukocytes. These factors are produced in the peripheral region to the photocoagulated area. The laser stimulates the production of adhesion molecules in the area around the shot and in the non photocoagulated area, which produces bearings and recruitment of leukocytes, secondary accumulation in the posterior pole and subsequent alteration of the hemato-retinal barrier (7).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 25 years, with a diagnosis of severe NPDR or PRD.
* Good pupil mydriasis (minimum 5mm) With clear media
* Patients without previous laser treatment or treatment with antiangiogenic drug.

Exclusion Criteria:

* Patients who do not accept informed consent.
* Patients with clinical macular Edema before treatment.
* Significant corneal opacity.
* Patients with other eye diseases that interfere with the studies required for the monitoring of patients.
* History of refractive surgery, glaucoma or ocular hypertension, intraocular inflammation, choroiditis multifocal, retinal detachment, optic neuropathy (4).
* Patients with tractional retinal detachment due to abundant fibrovascular

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Changes in a wave amplitude | 12 weeks
changes in b wave amplitude | 12 weeks
changes in ERG implicit time | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raul Velez-Montoya, MD, Principal Investigator — Asociaciòn para Evitar la Ceguera en Mèxico; Hugo Quiroz-Mercado, MD, Principal Investigator — Asociaciòn para Evitar la Ceguera en Mèxico; Virgilio Morales-Canton, MD, Principal Investigator — Asociaciòn para Evitar la Ceguera en Mèxico; Juan Manuel Jimenez-Sierra, MD, Principal Investigator — Asociaciòn para Evitar la Ceguera en Mèxico
Locations (1):
- Asociaciòn para Evitar la Ceguera en Mèxico, Mèxico, Mexico City, Mexico

REFERENCES:
- [Background] Blumenkranz MS, Yellachich D, Andersen DE, Wiltberger MW, Mordaunt D, Marcellino GR, Palanker D. Semiautomated patterned scanning laser for retinal photocoagulation. Retina. 2006 Mar;26(3):370-6. doi: 10.1097/00006982-200603000-00024. No abstract available. PMID 16508446
- [Background] Perlman I, Gdal-On M, Miller B, Zonis S. Retinal function of the diabetic retina after argon laser photocoagulation assessed electroretinographically. Br J Ophthalmol. 1985 Apr;69(4):240-6. doi: 10.1136/bjo.69.4.240. PMID 4039601
- [Background] Greenstein VC, Chen H, Hood DC, Holopigian K, Seiple W, Carr RE. Retinal function in diabetic macular edema after focal laser photocoagulation. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3655-64. PMID 11006264
- [Background] Varano M, Parisi V, Tedeschi M, Sciamanna M, Gallinaro G, Capaldo N, Catalano S, Pascarella A. Macular function after PDT in myopic maculopathy: psychophysical and electrophysiological evaluation. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1453-62. doi: 10.1167/iovs.04-0903. PMID 15790915
- [Background] Liang JC, Fishman GA, Huamonte FU, Anderson RJ. Comparative electroretinograms in argon laser and xenon arc panretinal photocoagulation. Br J Ophthalmol. 1983 Aug;67(8):520-5. doi: 10.1136/bjo.67.8.520. PMID 6683566
- [Background] Rema M, Sujatha P, Pradeepa R. Visual outcomes of pan-retinal photocoagulation in diabetic retinopathy at one-year follow-up and associated risk factors. Indian J Ophthalmol. 2005 Jun;53(2):93-9. doi: 10.4103/0301-4738.16171. PMID 15976463
- [Background] Nonaka A, Kiryu J, Tsujikawa A, Yamashiro K, Nishijima K, Kamizuru H, Ieki Y, Miyamoto K, Nishiwaki H, Honda Y, Ogura Y. Inflammatory response after scatter laser photocoagulation in nonphotocoagulated retina. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):1204-9. PMID 11923267